CLINICAL TRIAL: NCT00201955
Title: Rebamipide Ophthalmic Suspension in the Treatment of Dry Eye: A Multicenter, Phase 3, Randomized, Double-Masked, Placebo-Controlled, Parallel-Group, 26 Week Study
Brief Title: Study of Rebamipide Eye Drops to Treat Dry Eye
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 37E-03-201
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2006-11-02 (Estimated); Status verified 2006-10

CONDITIONS: Keratoconjunctivitis Sicca
Keywords: dry eye; keratoconjunctivitis sicca
MeSH Terms: conditions — Keratoconjunctivitis Sicca; Dry Eye Syndromes | interventions — rebamipide

INTERVENTIONS:
Drug: Rebamipide

SUMMARY:
The purpose of this study is to determine the potential safety and effectiveness of rebamipide eye drops, an investigational eye drop being developed for the treatment of keratoconjunctivitis sicca (dry eye).

DETAILED DESCRIPTION:
There is a need for effective therapy for dry eye that treats the underlying cause of the syndrome. The goal of this study is to assess the impact of rebamipide on dry eye symptoms.

ELIGIBILITY:
Inclusion Criteria:

* must have symptoms of dry eye for a minimum of 6 months
* must be able to sign and date an informed consent

Exclusion Criteria:

* presence of anterior segment disease
* glaucoma or ocular hypertension
* using Restasis
* use of topically instilled ocular medications during study
* use of contact lenses
* history of ocular surgery within 12 months
* females who are pregnant, breast feeding, or child-bearing potential and not willing to remain abstinent or use contraception
* presence of Stevens-Johnson syndrome
* any anticipated change in medication through-out study
* concurrent involvement in another study or previous receipt of this drug
* cannot be safely be weaned off of ocular medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 740
Dates: Start 2004-05; Study Completion 2006-07

PRIMARY OUTCOMES:
fluorescein corneal staining (FCS) total score at week 12 and the average primary ocular discomfort (POD) severity score at week 12

SECONDARY OUTCOMES:
fluorescein corneal staining (FCS) total score at week 26 and the average primary ocular discomfort (POD) severity score at week 26

CONTACTS AND LOCATIONS:
Locations (60):
- United States (60):
  - Harold Helms, MD, Birmingham, Alabama
  - Michael Bernstein, MD, Birmingham, Alabama
  - I Care! Eye Care!, Flagstaff, Arizona
  - Harvey and Bernice Jones Eye Institute, Little Rock, Arkansas
  - United Medical Research Institute, Inglewood, California
  - Benchmark Research, San Francisco, California
  - Southern California Clinical Research, Inc., San Marino, California
  - Colorado Eye Associates, PC, Colorado Springs, Colorado
  - Danbury Eye Physicians and Surgeons, P.C., Danbury, Connecticut
  - Florida Ophthalmic Institute, Gainesville, Florida
  - Florida Wellcare Alliance, L.C., Inverness, Florida
  - Shettle Eye Center, Largo, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Tukio Institute for Clinical Research, North Miami Beach, Florida
  - Magnolia Research Group, Inc., Ocala, Florida
  - Radiant Research - West Palm Beach, West Palm Beach, Florida
  - Vision Incorporated, Savannah, Georgia
  - Welborn Clinic, Evansville, Indiana
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Wichita Clinic, PA, Wichita, Kansas
  - Taustine Eye Center, Louisville, Kentucky
  - Bossier Optical, Inc., Bossier City, Louisiana
  - Stevenson Medical Surgical Eye Center, New Orleans, Louisiana
  - Family Eye Centers, New Orleans, Louisiana
  - Ophthalmic Research Associates, Inc., North Andover, Massachusetts
  - Minnesota Eye Associates, Minneapolis, Minnesota
  - Depremont Eye Specialists, Gulfport, Mississippi
  - Opthalmology Associates, Creve Coeur, Missouri
  - Clinical Research Laboratories, Piscataway, New Jersey
  - Ophthalmology Associates, Princeton, New Jersey
  - Eye Care Associates, Bethpage, New York
  - Ophthmalmic Consultants of Long Island, Lynbrook, New York
  - Mt. Sinai Medical Center School of Medicine, New York, New York
  - Rochester Ophthalmological Group, Rochester, New York
  - Ophthalmic Consultants of Long Island, Rockville Centre, New York
  - Ophthalmic Consultants of Long Island, Valley Stream, New York
  - Western Wake Eye Center, P.A., Cary, North Carolina
  - Southeast Clinical Research Associates, Charlotte, North Carolina
  - Horizon Eye Care - Clinical Research Dept., Charlotte, North Carolina
  - Cornerstone Research Care, High Point, North Carolina
  - Carolina Eye Associates, Southern Pines, North Carolina
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Comprehensive Opthalmology & Optical Services, Cleveland, Ohio
  - Bend Medical Clinic, Bend, Oregon
  - Medical Eye Center, Medford, Oregon
  - Valley Clinical Research Center, Easton, Pennsylvania
  - Philadelphia Eye Associates, Philadelphia, Pennsylvania
  - University of Pittsburg Eye and Ear Institute, Pittsburgh, Pennsylvania
  - Glaucome-Cataract Consultants, Pittsburgh, Pennsylvania
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Total Eye Care, P.A., Memphis, Tennessee
  - Corona Research Consultants, Inc., El Paso, Texas
  - The University of Texas Medical Branch, Galveston, Texas
  - Physician Research Network, Houston, Texas
  - Houston, Texas
  - Medical Center Ophthalmology, Houston, Texas
  - Houston Eye Associates, Houston, Texas
  - Sun Research Institute, San Antonio, Texas
  - Eye Clinic of South Texas, San Antonio, Texas
  - Advanced Healthcare Clinical Research Center, Milwaukee, Wisconsin